CLINICAL TRIAL: NCT03740412
Title: Intervention to Reduce Sedentary Time in Older Adults Undergoing Orthopaedic Surgery: a Feasibility Study (INTEREST)
Brief Title: Study to Reduce Sitting in Older Adults Undergoing Hip or Knee Replacements
Acronym: INTEREST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Birmingham (Other)
Collaborators: European Commission (Other); Dudley NHS Foundation Trust (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RG_17-169
Record Dates: First submitted 2017-12-04; First posted 2018-11-14 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Orthopedic Disorder; Arthropathy of Knee; Arthropathy of Hip; Sedentary Lifestyle; Physical Activity; Osteoarthritis
Keywords: sedentary; arthroplasty; osteoarthritis; older adults; elderly; old; elders; sitting; intervention
MeSH Terms: conditions — Musculoskeletal Diseases; Sedentary Behavior; Motor Activity; Osteoarthritis | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sedentary behaviour reduction (behaviour change techniques) (Experimental): Intervention group attending visits 1, 2, 3, 4, 5
  Interventions: Behavioral: Sedentary behaviour reduction using motivational interviewing, education, individualised feedback, goal-setting, self-monitoring, environmental modification, and supportive phone calls
- Usual care (No Intervention): Will receive usual orthopaedic care, attending visits 1, 4, 5

INTERVENTIONS:
Behavioral: Sedentary behaviour reduction using motivational interviewing, education, individualised feedback, goal-setting, self-monitoring, environmental modification, and supportive phone calls — The intervention has multiple components in order to reduce sedentary behaviour, namely: incorporating individualised feedback on sitting time, education about sedentary behaviour, individualised goal-setting and environmental modification according to each participant's own behavioural patterns and capabilities, motivational interviewing, and biweekly phone calls.
  Arms: Sedentary behaviour reduction (behaviour change techniques)

SUMMARY:
The aim of this study is to investigate the feasibility of an intervention to reduce sedentary behaviour in older adults waiting for hip and knee replacements. The study will be a randomised controlled trial design, including 2:1 randomisation into an intervention and usual care group respectively. A target of n=45 patients ≥60 years will be recruited from Russells Hall Hospital, Dudley, UK, approximately 8-10 weeks before surgery, assisted by research nurses. The variable-length intervention, informed by Self-Determination Theory (SDT), will be composed of multiple behaviour change techniques, namely motivational interviewing, individualised feedback on sedentariness, goal-setting, environmental modification, self-monitoring, and social support. Assessments will occur at baseline, 1 week pre-surgery, and 6 weeks post-surgery. The primary outcome will be the feasibility of the trial, assessed quantitatively using study statistics, and with mixed-methods assessment of acceptability, practicality, adaption, satisfaction, and safety via questionnaires given to participants. Exploratory outcomes will include physical function, cardiometabolic biomarkers, measurement of SDT constructs, and both objective and subjective measurement daily activity and sedentariness. The study will last up to 18 weeks per participant.

DETAILED DESCRIPTION:
The aim of this study is to investigate the feasibility of an intervention to reduce sedentary behaviour in n=45 older adults undergoing orthopaedic surgery, at Russells Hall Hospital, Dudley, Birmingham, UK. Recruitment will be via screening of surgery lists followed by direct contact with potentially eligible participants. The intervention is designed utilising Self Determination Theory. It is designed to have multiple components: incorporating individualised feedback on sitting time, education about sedentary behaviour, individualised goal-setting and environmental modification according to each participant's own behavioural patterns and capabilities, motivational interviewing, and biweekly phone calls.

Due to variation in surgery times, the intervention will be variable but can last up to 18 weeks. Each participant will undertake 3-5 visits depending on whether they are in the control group (n=3 visits) or intervention group (n=5 visits). The intervention group will undergo baseline assessments, two intervention meetings, pre-surgical assessments, and a 6-week post-surgical follow up. These visits will occur in different weeks for each participant due to the variability of surgery, however visit 2 will occur 1 week after visit 1. Visit 3 will occur shortly thereafter but may also be combined with visit 2. Visit 4 will occur the week prior to surgery, which is intended to be 6-10 weeks after baseline. Visit 5 occurs 6 weeks post-surgery, which should be 12-18 weeks post-baseline. The primary outcome measure will be feasibility, assessed quantitatively with study statistics. Secondary outcome will be mixed-methods assessment of feasibility via bespoke participant questionnaires. Exploratory outcomes will cover a number of mental and physical health variables, including blood measures to assess cardiometabolic biomarkers, as well as physical function using the short physical performance battery (SPPB). Surgical recovery will be assessed using the Oxford Hip/Knee score and the SPPB. The results of this feasibility study will serve to aid the design of a definitive trial of an intervention to reduce sedentary behaviour in this population.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged ≥60 years.
2. Listed for elective hip or knee surgery.
3. Capable of providing informed consent.
4. Regular access to a phone at pre-specified times.
5. Able to speak English.

Exclusion Criteria:

1. Neuromuscular impairments that preclude participating in physical activity, visual, hearing, or moderate/ severe cognitive impairments as indicated by the research nurse prior to recruitment.
2. Significant co-morbid disease that would pose a safety threat, affect blood measures significantly, or impair ability to participate such as coronary artery disease, severe hypertension, peripheral vascular disease, stroke, congestive heart failure, chronic obstructive pulmonary disease, insulin-dependent diabetes, psychiatric disease, renal disease, liver disease, or an active cancer other than skin cancer.
3. Working more than 2 days per week.
4. Unwillingness or inability to comply with the intervention.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-01-29 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2019-04-15 (Actual)

PRIMARY OUTCOMES:
Study uptake rates (as % of those approached who are randomised, recruitment rates (N/mth) | Assessed post-study-endpoint (up to month 18)
  Study uptake rates (as % of those approached who are randomised, recruitment rates (N/mth)
Intervention adherence to goals | Assessed post-study-endpoint (up to month 18)
  Self-recording by participants of goal achievement on a scale of 1-5, recorded each week for the first 6 weeks of the intervention in their goal-setting booklet.
Percentage of participants whose surgery is scheduled up to 2 weeks prior to the end of the intervention | Assessed post-study-endpoint (up to month 18)
  Percentage of participants whose surgery is scheduled up to 2 weeks prior to the end of the intervention
Percentage of participants whose surgery is scheduled up to three weeks after the end of the intervention | Assessed post-study-endpoint (up to month 18)
  Percentage of participants whose surgery is scheduled up to three weeks after the end of the intervention
Percentage of participants whose surgery is cancelled or delayed for too long | Assessed post-study-endpoint (up to month 18)
  Percentage of participants whose surgery is delayed beyond 3 weeks post-intervention
Retention rates (% of participants randomised who provide data at follow-up) | Assessed post-study-endpoint (up to month 18)
  Assessed by the number of participants who attend the follow-up visit (visit 5, 6 weeks post-surgery)
Acceptability of intervention for participants | Pre-surgery (visit 4, up to week 10), post-surgery (visit 5, up to week 18)
  Assessed by custom-made feasibility questionnaire which uses a number of closed and open questions. Closed questions include (Likert 1-5 scale):
  How easy was it to achieve your goals physically? How easy was it to achieve your goals mentally? Have you found taking part in the study burdensome?
Practicality of intervention for participants | Pre-surgery (visit 4, up to week 10), post-surgery (visit 5, up to week 18)
  Assessed by custom-made feasibility questionnaires, using both closed and open questions. Closed questions include (1-5 Likert scale):
  Could you have changed your goals to make them more achievable? Which part(s) of the intervention did you find most difficult?
Participant satisfaction with the study | Pre-surgery (visit 4, up to week 10), post-surgery (visit 5, up to week 18)
  Whether patients are satisfied, as assessed by feasibility questionnaires given at visit 4 (week prior to surgery) and visit 5 (week post-surgery). This included open and closed questions. Closed questions include (Likert scale 1-5):
  Which part(s) of the intervention did you find most enjoyable? How would you rate your overall satisfaction with the study? How likely would you be to suggest taking part in such a study to friends or family? How likely are you to continue working towards your goals in the future?
Patient perception of the safety of the study as assessed by questionnaire | Pre-surgery (visit 4, up to week 10), post-surgery (visit 5, up to week 18)
  Any change in patient safety as assessed by custom-made feasibility questionnaires. This includes closed and open questions. Closed questions include (Likert 1-3 scale):
  Do you feel that taking part in the study has exposed you to more pain? Do you feel that taking part in the study has exposed you to risk of physical harm?

SECONDARY OUTCOMES:
Short Physical Performance Battery (SPPB) | Baseline (visit 1, week 1), Pre-surgery (visit 4, up to week 10), post-surgery (visit 5, up to week 18)
  Short Physical Performance Battery (SPPB)
Sitting time | Baseline (visit 1, week 1), Pre-surgery (visit 4, up to week 10), post-surgery (visit 5, up to week 18)
  Assessed via activpal, mean minutes per day
Standing time | Baseline (visit 1, week 1), Pre-surgery (visit 4, up to week 10), post-surgery (visit 5, up to week 18)
  Assessed via activpal, mean minutes per day
Stepping time | Baseline (visit 1, week 1), Pre-surgery (visit 4, up to week 10), post-surgery (visit 5, up to week 18)
  Assessed via activpal, mean minutes per day
Sit-to-stand transitions | Baseline (visit 1, week 1), Pre-surgery (visit 4, up to week 10), post-surgery (visit 5, up to week 18)
  Assessed via activpal, n/day
Quantity of sedentary bouts >30 minutes | Baseline (visit 1, week 1), Pre-surgery (visit 4, up to week 10), post-surgery (visit 5, up to week 18)
  Assessed via activpal, n/day
Measure of Older Adults' Sedentary Time (MOST) | Baseline (visit 1, week 1), Pre-surgery (visit 4, up to week 10), post-surgery (visit 5, up to week 18)
  Measure of Older Adults' Sedentary Time (MOST)
EuroQol five dimensions questionnaire (EQ-5D) | Baseline (visit 1, week 1), Pre-surgery (visit 4, up to week 10), post-surgery (visit 5, up to week 18)
  EuroQol five dimensions questionnaire (EQ-5D) Assessed for each subscale (1-5 score on each); Mobility, Self-Care, Usual Activities, Pain, and Anxiety
EQ-VAS | Baseline (visit 1, week 1), Pre-surgery (visit 4, up to week 10), post-surgery (visit 5, up to week 18)
  Scale of overall perceived health on that day: scale 1-100 (100 is best, 0 is worst)
Oxford Hip/Knee Score | Baseline (visit 1, week 1), Pre-surgery (visit 4, up to week 10), post-surgery (visit 5, up to week 18)
  Oxford Hip/Knee Score. Reported as a scale from 0-48, where 0 is the most severe hip/knee osteoarthritis, and 48 is no indication of hip/knee osteoarthritis.
Basic Psychological Needs Scale | Baseline (visit 1, week 1), Pre-surgery (visit 4, up to week 10), post-surgery (visit 5, up to week 18)
  Three subscales: autonomy, relatedness, and competence. R equals reverse scoring. Max score for each is 49. Total score is not computed.
  Autonomy:
  1, 4(R), 8, 11(R), 14, 17, 20(R)
  Competence:
  3(R), 5, 10, 13, 15(R), 19(R)
  Relatedness:
  2, 6, 7(R), 9, 12, 16(R), 18(R), 21
International Physical Activity Questionnaire (IPAQ) Short Form | Baseline (visit 1, week 1), Pre-surgery (visit 4, up to week 10)
  The International Physical Activity Questionnaire (IPAQ) Short Form asks the amount of hours spent doing vigorous, moderate, and walking activities per day, and for how many days. It also asks for the average perceived sitting time per day.This gives a score for self-reported Vigorous Physical Activity, Moderate Physical Activity, Walking, and Sitting time.
Katz Activites of Daily Living | Baseline (visit 1, week 1), Pre-surgery (visit 4, up to week 10)
  Each item assess independence, in several domains, namely has a maximal overall score of 6 indicating maximal independence. The items are Bathing, Dressing, Toileting, Continence, Transferring (from bed to chair) and Feeding.
Body weight | Baseline (visit 1, week 1), Pre-surgery (visit 4, up to week 10), post-surgery (visit 5, up to week 18)
  KGs
Height | Baseline (visit 1, week 1)
  CMs
Body mass index | Baseline (visit 1, week 1), Pre-surgery (visit 4, up to week 10)
  kg/m2
Waist to hip ratio | Baseline (visit 1, week 1), Pre-surgery (visit 4, up to week 10)
  Waist to Hip Ratio (WHR) = Gw / Gh
Short Form Mini Nutritional Assessment (SF-MNA) | Baseline (visit 1, week 1)
  Short Form Mini Nutritional Assessment (SF-MNA). Gives a scale from 0-14, where 0 is most severely malnourished.
Albumin concentration | Baseline (visit 1, week 1), Pre-surgery (visit 4, up to week 10)
  Albumin
High Density Lipoprotein concentration | Baseline (visit 1, week 1), Pre-surgery (visit 4, up to week 10)
  High Density Lipoprotein
Low density lipoprotein concentration | Baseline (visit 1, week 1), Pre-surgery (visit 4, up to week 10)
  Low density lipoprotein
Triglyceride concentration | Baseline (visit 1, week 1), Pre-surgery (visit 4, up to week 10)
  Triglycerides
Vitamin D level | Baseline (visit 1, week 1), Pre-surgery (visit 4, up to week 10)
  Vitamin D
C-Reactive Protein concentration | Baseline (visit 1, week 1), Pre-surgery (visit 4, up to week 10)
  C-Reactive Protein
Interleukin 6 concentration | Baseline (visit 1, week 1), Pre-surgery (visit 4, up to week 10)
  Interleukin 6
Tumor Necrosis Factor Alpha concentration | Baseline (visit 1, week 1), Pre-surgery (visit 4, up to week 10)
  Tumor Necrosis Factor Alpha
Cortisol concentration | Baseline (visit 1, week 1), Pre-surgery (visit 4, up to week 10)
  Cortisol
Dehydroepiandrosterone sulfate (DHEAS) concentration | Baseline (visit 1, week 1), Pre-surgery (visit 4, up to week 10)
  Dehydroepiandrosterone sulfate
Transferrin concentration | Baseline (visit 1, week 1), Pre-surgery (visit 4, up to week 10)
  Transferrin

CONTACTS AND LOCATIONS:
Overall Officials: Justin Aunger, BA, Principal Investigator — Principal Investigator
Locations (1):
- Russells Hall Hospital, Dudley, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Aunger JA, Greaves CJ, Davis ET, Asamane EA, Whittaker AC, Greig CA. A novel behavioural INTErvention to REduce Sitting Time in older adults undergoing orthopaedic surgery (INTEREST): results of a randomised-controlled feasibility study. Aging Clin Exp Res. 2020 Dec;32(12):2565-2585. doi: 10.1007/s40520-020-01475-6. Epub 2020 Jan 23. PMID 31975288
- [Derived] Aunger JA, Greaves CJ, Davis ET, Greig CA. A novel behavioural INTErvention to REduce Sitting Time in older adults undergoing orthopaedic surgery (INTEREST): protocol for a randomised controlled feasibility study. Pilot Feasibility Stud. 2019 Apr 6;5:54. doi: 10.1186/s40814-019-0437-2. eCollection 2019. PMID 30997142